CLINICAL TRIAL: NCT01040689
Title: Randomised, Double-blind, Double-dummy, Placebo-controlled, 4-way Cross-over Study to Characterise the 24-hour Forced, Expiratory Volume After 1 Second (FEV1) Time Profiles of BI 1744 CL 5µg and 10µg (Oral Inhalation, Delivered by the Respimat® Inhaler) and Tiotropium Bromide 18µg (Oral Inhalation, Delivered by the HandiHaler®) After 6 Weeks of Treatment in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Characterization of 24 Hour Spirometry Profiles of Inhaled BI 1744 CL and Inhaled Tiotropium Bromide in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.39; 2009-014417-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

ARMS (4):
- Placebo (Placebo Comparator): olodaterol placebo and/or Tiotropium placebo inhaled once daily
  Interventions: Drug: Placebo (for olodaterol BI1744); Drug: Placebo (for Tiotropium)
- Olodaterol (BI1744) Low (Experimental): Low dose inhaled orally once daily from Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744) Low
- Olodaterol (BI1744) High (Experimental): High dose inhaled orally once daily from Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744) High
- Tiotropium 18 mcg (Active Comparator): 18mcg inhaled once daily from Handihaler
  Interventions: Drug: Tiotropium 18 mcg

INTERVENTIONS:
Drug: Olodaterol (BI1744) Low — Low dose inhaled orally once daily from Respimat inhaler
  Arms: Olodaterol (BI1744) Low
Drug: Placebo (for olodaterol BI1744) — Placebo (olodaterol low and high dose)delivered by Respimat
  Arms: Placebo
Drug: Placebo (for Tiotropium) — Placebo (Tiotropium 18 mcg) delivered by HandiHaler
  Arms: Placebo
Drug: Olodaterol (BI1744) High — High dose inhaled orally once daily from Respimat inhaler
  Arms: Olodaterol (BI1744) High
Drug: Tiotropium 18 mcg — 18mcg inhaled once daily from Handihaler
  Arms: Tiotropium 18 mcg

SUMMARY:
The study is intended to characterize the lung function profile of BI1744 in COPD patients where patients will perform pulmonary function tests at regular intervals for 24 hours at the end of a 6 week treatment period. Each patient will receive all four treatments.

ELIGIBILITY:
Inclusion criteria:

* Patients willing to participate with confirmed diagnosis of COPD
* 40 years of age or older
* having a 10 pack year smoking history
* able to perform serial pulmonary function tests
* able to use both a Dry powder inhaler (DPI) and Respimat device

Exclusion criteria:

* Significant other disease
* clinically relevant abnormal hematology, chemistry, or urinalysis
* history of asthma
* diagnosis of thyrotoxicosis
* paroxysmal tachycardia related to beta agonists
* history of MI within 1 year, cardiac arrhythmia, hospitalization for heart failure within 1 year
* active tuberculosis, cystic fibrosis, clinically evident bronchiectasis
* significant alcohol or drug abuse
* pulmonary resection
* taking oral beta adrenergics
* taking unstable oral steroids
* daytime oxygen
* enrolled in rehabilitation program
* enrolled in another study or taking investigational products
* pregnant or nursing women, women of child bearing potential not willing to use two methods of birth control
* those who are not willing to comply with pulmonary medication washouts

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- Belgium (3):
  - 1222.39.32003 Boehringer Ingelheim Investigational Site, Genk
  - 1222.39.32001 Boehringer Ingelheim Investigational Site, Ghent
  - 1222.39.32002 Boehringer Ingelheim Investigational Site, Hasselt
- Denmark (3):
  - 1222.39.45001 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1222.39.45003 Boehringer Ingelheim Investigational Site, Kolding
  - 1222.39.45002 Boehringer Ingelheim Investigational Site, Odense C
- Germany (3):
  - 1222.39.49391 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.39.49392 Boehringer Ingelheim Investigational Site, Hamburg
  - 1222.39.49393 Boehringer Ingelheim Investigational Site, Mannheim
- Hungary (6):
  - 1222.39.36006 Boehringer Ingelheim Investigational Site, Deszk
  - 1222.39.36004 Boehringer Ingelheim Investigational Site, Farkasgyepü
  - 1222.39.36005 Boehringer Ingelheim Investigational Site, Pécs
  - 1222.39.36003 Boehringer Ingelheim Investigational Site, Szarvas
  - 1222.39.36001 Boehringer Ingelheim Investigational Site, Szeged
  - 1222.39.36002 Boehringer Ingelheim Investigational Site, Törökbálint

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. The duration of each treatment period was 6 weeks with a 3 week washout period between treatments.
Groups:
- Placebo / Tio 18mcg / Olo 10mcg / Olo 5mcg: Patients were administered placebo in the first period, Tiotropium 18 mcg qd in the second period, Olodaterol 10 mcg qd in the third period and Olodaterol 5 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Olo 5mcg / Olo 10mcg / Tio 18mcg / Placebo: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 10 mcg qd in the second period, Tiotropium 18 mcg qd in the third period and placebo in the fourth period. Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Olo 10mcg / Placebo / Olo 5mcg / Tio 18mcg: Patients were administered Olodaterol 10 mcg qd in the first period, placebo in the second period, Olodaterol 5 mcg qd in the third period and Tiotropium 18 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Tio 18mcg / Olo 5mcg / Placebo / Olo 10mcg: Patients were administered Tiotropium 18 mcg qd in the first period, Olodaterol 5 mcg qd in the second period, placebo in the third period and Olodaterol 10 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
Period: Overall Study
Arm/Group | Placebo / Tio 18mcg / Olo 10mcg / Olo 5mcg | Olo 5mcg / Olo 10mcg / Tio 18mcg / Placebo | Olo 10mcg / Placebo / Olo 5mcg / Tio 18mcg | Tio 18mcg / Olo 5mcg / Placebo / Olo 10mcg
Started | 27 | 27 | 27 | 27
Completed | 24 | 25 | 23 | 23
Not Completed | 3 | 2 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 2 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Other reasons not listed above | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. 108 patients were assigned randomly to one of 4 treatment sequences in which they received each of 4 treatments, two doses (5 microgram (mcg) or 10 mcg) of Olodaterol (Olo) once daily (qd) delivered via the Respimat inhaler or Tiotropium (Tio) 18 mcg once daily (qd) delivered via the HandiHaler or equivalent placebo. The duration of each treatment period was 6 weeks with a 3 week washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 83

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit for the first period, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of the first treatment period (study baseline) and -30 min (zero time), 30 min, 60 min, 2 hour (h) , 3 h, 4 h, 6 h, 8 h, 10 h, 12 h relative to am dose after six weeks of treatment
Population: Full analysis set (FAS). FAS is defined as all patients with baseline (pre-dose) data and any evaluable post-dosing data for either co-primary endpoint from the same treatment period. FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler or Handihaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Tio 18 mcg qd: Tiotropium (Tio) 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.054 (0.020) | 0.131 (0.020) | 0.152 (0.020) | 0.119 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate; Mean Difference (Final Values) = 0.185, 95% CI [0.145 to 0.224], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI [0.167 to 0.246], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.133 to 0.212], Standard Error of Mean 0.020 — Tio 18 mcg qd minus Placebo

2. Primary Outcome: FEV1 Area Under Curve 12-24h (AUC 12-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit for the first period, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of the first treatment period (study baseline) and 12 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Tio 18 mcg qd: Tiotropium 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.095 (0.021) | 0.036 (0.021) | 0.082 (0.021) | 0.027 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.131, 95% CI [0.090 to 0.173], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.136 to 0.219], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI [0.081 to 0.164], Standard Error of Mean 0.021 — Tio 18 mcg qd minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 h (AUC 0-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the first visit of the first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h, 4 h, 6h, 8h, 10h, 12 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.075 (0.020) | 0.083 (0.020) | 0.117 (0.020) | 0.073 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.158, 95% CI [0.121 to 0.196], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.155 to 0.230], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.148, 95% CI [0.110 to 0.185], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After First Dose of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of the first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-3h was calculated from 0-3hours post-dose using the trapezoidal rule, divided by the observation time (3 h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose of the first period (study baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to the first dose of treatment period
Population: FAS including all patients with evaluable data after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 101 | 101 | 100 | 98
Liter | -0.021 (0.017) | 0.161 (0.017) | 0.191 (0.017) | 0.111 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.147 to 0.216], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.178 to 0.247], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.132, 95% CI [0.097 to 0.167], Standard Error of Mean 0.018 — Tio 18 mcg qd minus Placebo

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After Six Weeks of Treatment
Description: as for outcome 4
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to the last dose of treatment after six weeks of treatment.
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.045 (0.019) | 0.161 (0.019) | 0.170 (0.019) | 0.137 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.206, 95% CI [0.170 to 0.243], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.215, 95% CI [0.179 to 0.252], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.146 to 0.219], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

6. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of first treatment period. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after the first dose of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and first day of dosing
Population: FAS including all patients with evaluable data after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 101 | 101 | 100 | 98
Liter | 0.040 (0.018) | 0.253 (0.018) | 0.279 (0.018) | 0.201 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.177 to 0.249], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.239, 95% CI [0.203 to 0.275], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.125 to 0.197], Standard Error of Mean 0.018 — Tio 18 mcg qd minus Placebo

7. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of first treatment period. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after the last dose after six weeks of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | 0.019 (0.022) | 0.232 (0.022) | 0.253 (0.022) | 0.220 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.168 to 0.258], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.234, 95% CI [0.189 to 0.279], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.201, 95% CI [0.156 to 0.246], Standard Error of Mean 0.023 — Tio 18 mcg qd minus Placebo

8. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline trough FEV1 was defined as the mean of the available pre-dose trough FEV1 values prior to first dose of first treatment period. Trough values were the mean of values obtained 23 hours and 23h 50min post the last dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.043 (0.020) | 0.090 (0.020) | 0.104 (0.020) | 0.054 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.133, 95% CI [0.096 to 0.170], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.110 to 0.184], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.060 to 0.134], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

9. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose in first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of the first treatment period (study baseline) and -30 min (zero time), 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12h relative to last dose after six weeks of treatment.
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.110 (0.038) | 0.172 (0.038) | 0.192 (0.038) | 0.166 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.282, 95% CI [0.216 to 0.348], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.303, 95% CI [0.237 to 0.368], Standard Error of Mean 0.033 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.276, 95% CI [0.210 to 0.342], Standard Error of Mean 0.034 — Tio 18 mcg qd minus Placebo

10. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose of first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 h and 10 min prior to dose on the first day of the first treatment period (study baseline) and 12 h, 22 h, 23 h, and 23 h 50 min relative to last dose after six weeks of treatment
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.166 (0.039) | 0.030 (0.039) | 0.086 (0.039) | 0.018 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.196, 95% CI [0.131 to 0.262], Standard Error of Mean 0.033 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.252, 95% CI [0.187 to 0.318], Standard Error of Mean 0.033 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.184, 95% CI [0.118 to 0.249], Standard Error of Mean 0.033 — Tio 18 mcg qd minus Placebo

11. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose in first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h, 4 h, 6h, 8h, 10h, 12 h, 22 h, 23 h, and 23 h 50 min relative to last dose after six weeks of treatment.
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.138 (0.037) | 0.101 (0.037) | 0.139 (0.037) | 0.091 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.240, 95% CI [0.178 to 0.301], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.278, 95% CI [0.216 to 0.339], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.230, 95% CI [0.168 to 0.291], Standard Error of Mean 0.031 — Tio 18 mcg qd minus Placebo

12. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose in the first treatment period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-3h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of the treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h relative to first dose of treatment
Population: FAS including all patients with evaluable data after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 101 | 101 | 100 | 98
Liter | -0.024 (0.037) | 0.244 (0.037) | 0.288 (0.037) | 0.191 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.268, 95% CI [0.207 to 0.330], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.312, 95% CI [0.251 to 0.374], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.215, 95% CI [0.153 to 0.277], Standard Error of Mean 0.031 — Tio 18 mcg qd minus Placebo

13. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response
Description: as for outcome 12
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h relative to last dose after six weeks of treatment.
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.083 (0.040) | 0.234 (0.040) | 0.235 (0.040) | 0.219 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.317, 95% CI [0.246 to 0.388], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.318, 95% CI [0.247 to 0.388], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.302, 95% CI [0.231 to 0.373], Standard Error of Mean 0.036 — Tio 18 mcg qd minus Placebo

14. Secondary Outcome: Peak FVC (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FVC was defined as the mean of the available pre-dose peak FVC values prior to first dose in first treatment period. Peak FVC (0-3h) was obtained within 0 - 3 hours after the last dose of study drug after 6 weeks of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | 0.086 (0.043) | 0.386 (0.043) | 0.383 (0.043) | 0.381 (0.043)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.300, 95% CI [0.222 to 0.378], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.297, 95% CI [0.220 to 0.375], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.295, 95% CI [0.217 to 0.373], Standard Error of Mean 0.040 — Tio 18 mcg qd minus Placebo

15. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline trough FVC was defined as the mean of the available pre-dose trough FVC values prior to first dose in first treatment period. Trough values were mean of the values obtained 23 h and 23 h 50 min after the last dose of study drug after six weeks of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 99 | 100 | 99 | 99
Liter | -0.082 (0.041) | 0.103 (0.041) | 0.130 (0.041) | 0.046 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.185, 95% CI [0.115 to 0.255], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.212, 95% CI [0.143 to 0.282], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI [0.059 to 0.199], Standard Error of Mean 0.036 — Tio 18 mcg qd minus Placebo

16. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 6 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Tiotropium (Tio) 18 mcg qd: Tiotropium (Tio) 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Tiotropium (Tio) 18 mcg qd
Number analyzed (Participants) | 102 | 101 | 101 | 101
percentage of participants
  Palpitations | 0.0 | 0.0 | 1.0 | 0.0
  Investigations | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Tiotropium (Tio) 18 mcg qd
Serious Adverse Events (participants affected / at risk) | 5/102 | 1/101 | 0/101 | 5/101
Other Adverse Events (participants affected / at risk) | 12/102 | 14/101 | 6/101 | 10/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | Olo 5 mcg (N=101) | Olo 10 mcg (N=101) | Tiotropium (Tio) 18 mcg qd (N=101)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | Olo 5 mcg (N=101) | Olo 10 mcg (N=101) | Tiotropium (Tio) 18 mcg qd (N=101)
Nasopharyngitis (Infections and infestations) | 8 | 6 | 4 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication